CLINICAL TRIAL: NCT02749370
Title: Open Label Study to Evaluate the Efficacy of Etanercept Treatment in Subjects With Moderate to Severe Plaque Psoriasis Who Have Failed Therapy With Apremilast
Brief Title: Study to Evaluate the Efficacy of Etanercept Treatment in Adults Who Failed Therapy With Apremilast
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150252
Record Dates: First submitted 2016-03-14; First posted 2016-04-25 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental): Participants received etanercept 50 mg subcutaneously twice weekly for 12 weeks followed by 50 mg once weekly for an additional 12 weeks.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Administered subcutaneously twice weekly for 12 weeks then once weekly for an additional 12 weeks.
  Other Names: Enbrel

SUMMARY:
To evaluate the efficacy of etanercept in adults with moderate to severe plaque psoriasis who have failed therapy with apremilast (Otezla).

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, phase 4, estimation study in adults with plaque psoriasis (PsO) who have failed apremilast. The study will consist of a screening period of up to 45 days, a 24-week treatment period with study visits every 4 weeks, and a 30-day follow-up period for safety. Etanercept dosing will follow the recommended label dosing for adults with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study specific activities/procedures
* Male or female subject is ≥ 18 years of age at time of screening
* Subject is a candidate for systemic therapy or phototherapy in the opinion of the investigator
* Subject has moderate to severe plaque psoriasis (PsO) with involved body surface area (BSA) ≥ 10%, psoriasis area and severity index (PASI) ≥ 10 and static physician's global assessment (sPGA) ≥ 3 at screening and baseline
* Subject is currently receiving treatment with apremilast for moderate to severe plaque PsO or subject has discontinued treatment with apremilast for PsO within the past 3 months prior to screening
* Subject has failed therapy with apremilast for moderate to severe plaque PsO defined as either (1) failure to achieve adequate clinical response in the opinion of the investigator, (2) loss of adequate clinical response in the opinion of the investigator or (3) intolerability to apremilast in the opinion of the investigator
* Subject has received at least 4 weeks of apremilast treatment for moderate to severe plaque PsO (this only applies for subjects who are qualifying by failure to achieve adequate clinical response or loss of adequate clinical response, this does not apply for subjects who are qualifying by intolerability to apremilast)
* Subject has not had significant known weight increase or decrease (≥ 10%) during apremilast treatment
* Subject is < 264 lbs at screening and baseline -Subject has a negative test for hepatitis B surface antigen, hepatitis B core antibody and hepatitis C antibody
* Subject has no known history of tuberculosis.

Exclusion Criteria:

Skin disease related

-Subject has active erythrodermic, pustular, guttate psoriasis, or medication induced psoriasis, or other skin conditions at the time of the screening visit (for example, eczema) that would interfere with evaluations of the effect of investigational product on PsO.

Other Medical Conditions

* Subject has one or more significant concurrent medical conditions per investigator judgment, including the following
* Poorly controlled diabetes
* Chronic kidney disease stage IIIb, IV, or V
* Symptomatic heart failure (New York Heart Association class II, III, or IV)
* Myocardial infarction or unstable angina pectoris within the past 12 months prior to randomization
* Uncontrolled hypertension
* Severe chronic pulmonary disease (eg, requiring oxygen therapy)
* Multiple sclerosis or any other demyelinating disease
* Liver disease
* Anemia
* Major chronic inflammatory disease or connective tissue disease other than psoriasis and/or psoriatic arthritis (for example, systemic lupus erythematosus with the exception of secondary Sjogren's syndrome)
* Subject has active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma, Merkel cell carcinoma or history of cancer (other than fully resected and surgically cured cutaneous basal cell and squamous cell carcinoma) within 5 years before the first dose of investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- United States (22):
  - Research Site, Scottsdale, Arizona
  - Research Site, Beverly Hills, California
  - Research Site, Fountain Valley, California
  - Research Site, Newport Beach, California
  - Research Site, San Ramon, California
  - Research Site, Santa Monica, California
  - Research Site, Coral Gables, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Macon, Georgia
  - Research Site, Louisville, Kentucky
  - Research Site, Rockville, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Clarkston, Michigan
  - Research Site, Fort Gratiot, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Henderson, Nevada
  - Research Site, East Windsor, New Jersey
  - Research Site, Verona, New Jersey
  - Research Site, New York, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas

REFERENCES:
- [Background] Bagel J, Samad AS, Stolshek BS, Aras GA, Chung JB, Kricorian G, Kircik LH. Open-Label Study to Evaluate the Efficacy of Etanercept Treatment in Subjects With Moderate to Severe Plaque Psoriasis Who Have Failed Therapy With Apremilast. J Drugs Dermatol. 2018 Oct 1;17(10):1078-1082. PMID 30365588
- [Background] Bagel J, Stolshek BS, Yang Y, Kricorian G, Kircik LH. Evaluation of Patient-Reported Outcomes With Etanercept in Moderate to Severe Plaque Psoriasis Patients After Therapy With Apremilast. J Drugs Dermatol. 2020 Apr 1;19(4):378-383. doi: 10.36849/JDD.2020.4910. PMID 32272514
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 22 centers in the United States from 18 May 2016 to 06 December 2017.
Period: Overall Study
Arm/Group | Etanercept
Started | 80
Completed | 66
Not Completed | 14
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (14.8)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 63
  ≥ 65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 11
  Black or African American | 2
  Native Hawaiian or Other Pacific Islander | 0
  White | 60
  Other | 3
Psoriasis Area Severity Index (PASI) Score [Mean (Standard Deviation); unit: units on a scale] — The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0 to 72, with higher scores indicating greater severity and/or more extensive psoriasis.
  units on a scale | 16.4 (6.5)
Percent of Body Surface Area (BSA) Involved in Psoriasis [Mean (Standard Deviation); unit: Percentage of BSA] — A measurement of psoriasis involvement, given as the physician's assessment of the percentage of the participant's total body surface area involved with psoriasis.
  Percentage of BSA | 16.4 (10.5)
Static Physician Global Assessment (sPGA) of Psoriasis [Count of Participants; unit: Participants] — A physician's global assessment of the participant's psoriasis based on the severity of induration, scaling, and erythema. The sPGA of psoriasis is a 6-point scale ranging from 0 (clear) to 5 (very severe).
  Participants
    0 = Clear | 0
    1 = Almost clear | 0
    2 = Mild | 0
    3 = Moderate | 51
    4 = Severe | 28
    5 = Very Severe | 1
Dermatology Life Quality Index (DLQI) [Mean (Standard Deviation); unit: units on a scale] — The DLQI is a 10-item skin disease-specific instrument to evaluate impact of skin disease on health-related quality of life. Items rated on a 4-point Likert scale were summed to create a DLQI total score ranging from 0 (best possible score) to 30 (worst possible score). Total scores of the DLQI are interpreted as 0 to 1 = no effect at all on patient's life, 2 to 5 = small effect on patient's life, 6 to 10 = moderate effect on patient's life, 11 to 20 = very large effect on patient¡'s life, 21 to 30 = extremely large effect on patient¡'s life.
  units on a scale | 12.5 (7.4)
Psoriasis Symptom Inventory (PSI) [Mean (Standard Deviation); unit: units on a scale] — Participants rated the severity of their psoriasis signs and symptoms on an 8-item questionnaire (itch, redness, scaling, burning, stinging, cracking, flaking, pain) based on the past 7 days. Each item was scored on a 5-point scale from 0 (not at all severe) to 4 (very severe). The total score was calculated as the sum of the 8 responses, and ranges from 0 to 32. Each component score ranges from 0 to 4. Higher total score and component scores indicate more severe psoriasis.
  units on a scale
    Total score | 16.6 (6.6)
    Itch from psoriasis | 2.5 (1.0)
    Redness of skin lesions | 2.6 (0.9)
    Scaling of skin lesions | 2.6 (0.8)
    Burning of skin lesions | 1.4 (1.2)
    Stinging of skin lesions | 1.5 (1.2)
    Cracking of skin lesions | 2.0 (1.0)
    Flaking of skin lesions | 2.5 (1.9)
    Pain from skin lesions | 1.5 (1.1)
Patient Assessment of Treatment Satisfaction [Count of Participants; unit: Participants] — Participants indicated their level of satisfaction with the medication's control of psoriasis on a scale from "very dissatisfied" to "very satisfied".
  Participants
    Very dissatisfied | 33
    Dissatisfied | 13
    Neither satisfied nor dissatisfied | 30
    Satisfied | 4
    Very satisfied | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a PASI 75 Response at Week 12
Description: A PASI 75 response is a 75% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0 to 72, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and week 12
Population: Participants who received at least 1 dose of etanercept during the study and with at least 1 post-baseline PASI value. Last observation carried forward (LOCF) imputation was used for participants with missing data at week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 77
percentage of participants | 41.6 [30.4 to 53.4]

2. Secondary Outcome: Percentage of Participants With a PASI 75 Response at Each Visit
Description: as for outcome 1
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: Participants who received at least 1 dose of etanercept during the study and with at least 1 post-baseline PASI value. Last observation carried forward (LOCF) imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 77
percentage of participants
  Week 4: number analyzed (Participants) | 76
  Week 4 | 6.6 [2.2 to 14.7]
  Week 8 | 23.4 [14.5 to 34.4]
  Week 12 | 41.6 [30.4 to 53.4]
  Week 16 | 42.9 [31.6 to 54.6]
  Week 20 | 42.9 [31.6 to 54.6]
  Week 24 | 45.5 [34.1 to 57.2]

3. Secondary Outcome: Percentage of Participants With a PASI 50 Response at Each Visit
Description: A PASI 50 response is a 50% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0 to 72, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 77
percentage of participants
  Week 4: number analyzed (Participants) | 76
  Week 4 | 23.7 [14.7 to 34.8]
  Week 8 | 50.6 [39.0 to 62.2]
  Week 12 | 70.1 [58.6 to 80.0]
  Week 16 | 68.8 [57.3 to 78.9]
  Week 20 | 74.0 [62.8 to 83.4]
  Week 24 | 62.3 [50.6 to 73.1]

4. Secondary Outcome: Percentage of Participants With a PASI 90 Response at Each Visit
Description: A PASI 90 response is a 90% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0 to 72, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 77
percentage of participants
  Week 4: number analyzed (Participants) | 76
  Week 4 | 1.3 [0.0 to 7.1]
  Week 8 | 6.5 [2.1 to 14.5]
  Week 12 | 13.0 [6.4 to 22.6]
  Week 16 | 16.9 [9.3 to 27.1]
  Week 20 | 23.4 [14.5 to 34.4]
  Week 24 | 22.1 [13.4 to 33.0]

5. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI)
Description: The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0 to 72, with higher scores indicating greater severity and/or more extensive psoriasis.
  Percent change from baseline was calculated as (Baseline Value - Post-baseline Value) / Baseline Value * 100, hence a positive value indicates improvement.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 77
percent change
  Week 4: number analyzed (Participants) | 76
  Week 4 | 22.03 (33.58)
  Week 8 | 43.51 (40.53)
  Week 12 | 55.47 (48.16)
  Week 16 | 57.41 (40.79)
  Week 20 | 60.42 (39.12)
  Week 24 | 57.67 (40.20)

6. Secondary Outcome: Percentage of Participants With an sPGA Score of 0 (Clear) or 1 (Almost Clear) at Each Visit
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). A sPGA response is defined as a sPGA value of clear (score 0) or almost clear (score 1).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: Participants who received at least 1 dose of etanercept during the study and with at least 1 post-baseline sPGA value. Last observation carried forward (LOCF) imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 77
percentage of participants
  Week 4: number analyzed (Participants) | 76
  Week 4 | 3.9 [0.8 to 11.1]
  Week 8 | 15.6 [8.3 to 25.6]
  Week 12 | 23.4 [14.5 to 34.4]
  Week 16 | 28.6 [18.8 to 40.0]
  Week 20 | 29.9 [20.0 to 41.4]
  Week 24 | 33.8 [23.4 to 45.4]

7. Secondary Outcome: Percentage of Participants With an sPGA Score of 0, 1 or 2 at Each Visit
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). The percentage of participants with a score of 0 (clear), 1 (almost clear) or 2 (mild) is reported.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 77
percentage of participants
  Week 4: number analyzed (Participants) | 76
  Week 4 | 21.1 [12.5 to 31.9]
  Week 8 | 55.8 [44.1 to 67.2]
  Week 12 | 62.3 [50.6 to 73.1]
  Week 16 | 59.7 [47.9 to 70.8]
  Week 20 | 55.8 [44.1 to 67.2]
  Week 24 | 57.1 [45.4 to 68.4]

8. Secondary Outcome: Static Physician Global Assessment (sPGA) at Each Visit
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 77
units on a scale
  Week 4: number analyzed (Participants) | 76
  Week 4 | 2.9 (0.7)
  Week 8 | 2.4 (0.9)
  Week 12 | 2.2 (1.0)
  Week 16 | 2.2 (1.1)
  Week 20 | 2.2 (1.1)
  Week 24 | 2.2 (1.2)

9. Secondary Outcome: Percentage of Participants With at Least a 1 Grade Improvement in sPGA From Baseline
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). The percentage of participants with an improvement from baseline of ≥ 1 grade is reported.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 77
percentage of participants
  Week 4: number analyzed (Participants) | 76
  Week 4 | 40.8 [29.6 to 52.7]
  Week 8 | 70.1 [58.6 to 80.0]
  Week 12 | 75.3 [64.2 to 84.4]
  Week 16 | 72.7 [61.4 to 82.3]
  Week 20 | 74.0 [62.8 to 83.4]
  Week 24 | 74.0 [62.8 to 83.4]

10. Secondary Outcome: Percentage of Participants With at Least a 2 Grade Improvement in sPGA From Baseline
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). The percentage of participants with an improvement from baseline of ≥ 2 grades is reported.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: Participants who received at least 1 dose of etanercept during the study and with at least I post-baseline sPGA value. Last observation carried forward (LOCF) imputation was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 77
percentage of participants
  Week 4: number analyzed (Participants) | 76
  Week 4 | 7.9 [3.0 to 16.4]
  Week 8 | 31.2 [21.1 to 42.7]
  Week 12 | 32.5 [22.2 to 44.1]
  Week 16 | 37.7 [26.9 to 49.4]
  Week 20 | 36.4 [25.7 to 48.1]
  Week 24 | 39.0 [28.0 to 50.8]

11. Secondary Outcome: Percent Change From Baseline in the Percentage of Body Surface Area (BSA) Involved With Psoriasis at Each Visit
Description: A measurement of psoriasis involvement, given as the physician's assessment of the percentage of the participant's total body surface area (BSA) involved with psoriasis. The percent of BSA affected was estimated by assuming that the participant's palm, excluding the fingers and thumb, represented roughly 1% of the body's surface. Percent change from baseline was calculated as (Baseline Value - Post-baseline Value) / Baseline Value * 100, hence a positive value indicates improvement.
Time Frame: Baseline and weeks 4, 8, 12, 16, 20, and 24
Population: Participants who received at least 1 dose of etanercept during the study and with at least 1 post-baseline value. Last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 77
percent change
  Week 4: number analyzed (Participants) | 76
  Week 4 | 13.47 (24.63)
  Week 8 | 31.03 (37.52)
  Week 12 | 44.49 (40.29)
  Week 16 | 48.26 (39.80)
  Week 20 | 49.97 (40.15)
  Week 24 | 46.89 (42.70)

12. Secondary Outcome: Psoriasis Symptom Inventory (PSI) Total Score at Each Visit
Description: Participants rated the severity of their psoriasis signs and symptoms on an 8-item questionnaire (itch, redness, scaling, burning, stinging, cracking, flaking, pain) based on the past 7 days. Each item was scored on a 5-point scale from 0 (not at all severe) to 4 (very severe). The total score is the sum of the 8 responses, and ranges from 0 to 32. Higher scores indicate more severe psoriasis.
Time Frame: Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 77
units on a scale
  Week 1: number analyzed (Participants) | 74
  Week 1 | 14.7 (7.1)
  Week 2: number analyzed (Participants) | 74
  Week 2 | 13.7 (6.5)
  Week 3: number analyzed (Participants) | 74
  Week 3 | 12.1 (6.1)
  Week 4 | 11.7 (6.6)
  Week 8 | 10.0 (5.9)
  Week 12 | 8.8 (6.4)
  Week 16 | 10.1 (7.6)
  Week 20 | 9.9 (7.8)
  Week 24 | 9.6 (7.7)

13. Secondary Outcome: PSI "Itch From Psoriasis" Component Score at Each Visit
Description: Participants rated the severity of their psoriasis signs and symptoms on an 8-item questionnaire (itch, redness, scaling, burning, stinging, cracking, flaking, pain) based on the past 7 days. Each item was scored on a 5-point scale from 0 (not at all severe) to 4 (very severe).
Time Frame: Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 77
units on a scale
  Week 1: number analyzed (Participants) | 74
  Week 1 | 2.2 (1.0)
  Week 2: number analyzed (Participants) | 74
  Week 2 | 2.0 (0.9)
  Week 3: number analyzed (Participants) | 74
  Week 3 | 1.9 (0.8)
  Week 4 | 1.8 (0.9)
  Week 8 | 1.5 (0.9)
  Week 12 | 1.3 (0.9)
  Week 16 | 1.5 (1.0)
  Week 20 | 1.5 (1.1)
  Week 24 | 1.5 (1.0)

14. Secondary Outcome: PSI "Redness of Skin Lesions" Component Score at Each Visit
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 77
units on a scale
  Week 1: number analyzed (Participants) | 74
  Week 1 | 2.4 (0.9)
  Week 2: number analyzed (Participants) | 74
  Week 2 | 2.2 (0.9)
  Week 3: number analyzed (Participants) | 74
  Week 3 | 2.0 (0.8)
  Week 4 | 1.8 (0.9)
  Week 8 | 1.7 (0.9)
  Week 12 | 1.5 (1.0)
  Week 16 | 1.7 (1.1)
  Week 20 | 1.5 (1.1)
  Week 24 | 1.5 (1.1)

15. Secondary Outcome: PSI "Scaling of Skin Lesions" Component Score at Each Visit
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 77
units on a scale
  Week 1: number analyzed (Participants) | 74
  Week 1 | 2.3 (1.0)
  Week 2: number analyzed (Participants) | 74
  Week 2 | 2.1 (1.1)
  Week 3: number analyzed (Participants) | 74
  Week 3 | 1.9 (0.9)
  Week 4 | 1.9 (0.9)
  Week 8 | 1.6 (0.9)
  Week 12 | 1.5 (0.9)
  Week 16 | 1.6 (1.0)
  Week 20 | 1.6 (1.1)
  Week 24 | 1.4 (1.1)

16. Secondary Outcome: PSI "Burning of Skin Lesions" Component Score at Each Visit
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 77
units on a scale
  Week 1: number analyzed (Participants) | 74
  Week 1 | 1.3 (1.1)
  Week 2: number analyzed (Participants) | 74
  Week 2 | 1.2 (1.1)
  Week 3: number analyzed (Participants) | 74
  Week 3 | 1.0 (1.0)
  Week 4 | 1.0 (1.0)
  Week 8 | 0.8 (0.9)
  Week 12 | 0.8 (1.0)
  Week 16 | 0.9 (1.1)
  Week 20 | 0.9 (1.1)
  Week 24 | 0.9 (1.1)

17. Secondary Outcome: PSI "Stinging of Skin Lesions" Component Score at Each Visit
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 77
units on a scale
  Week 1: number analyzed (Participants) | 74
  Week 1 | 1.2 (1.2)
  Week 2: number analyzed (Participants) | 74
  Week 2 | 1.1 (1.0)
  Week 3: number analyzed (Participants) | 74
  Week 3 | 1.0 (1.0)
  Week 4 | 1.0 (1.1)
  Week 8 | 0.8 (0.9)
  Week 12 | 0.7 (0.9)
  Week 16 | 0.9 (1.1)
  Week 20 | 0.9 (1.1)
  Week 24 | 0.8 (1.1)

18. Secondary Outcome: PSI "Cracking of Skin Lesions" Component Score at Each Visit
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 77
units on a scale
  Week 1: number analyzed (Participants) | 74
  Week 1 | 1.9 (1.1)
  Week 2: number analyzed (Participants) | 74
  Week 2 | 1.7 (1.0)
  Week 3: number analyzed (Participants) | 74
  Week 3 | 1.6 (1.0)
  Week 4 | 1.4 (1.1)
  Week 8 | 1.2 (1.0)
  Week 12 | 1.1 (1.0)
  Week 16 | 1.2 (1.0)
  Week 20 | 1.2 (1.1)
  Week 24 | 1.2 (1.1)

19. Secondary Outcome: PSI "Flaking of Skin Lesions" Component Score at Each Visit
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 77
units on a scale
  Week 1: number analyzed (Participants) | 74
  Week 1 | 2.2 (0.9)
  Week 2: number analyzed (Participants) | 74
  Week 2 | 2.1 (0.9)
  Week 3: number analyzed (Participants) | 74
  Week 3 | 1.8 (0.9)
  Week 4 | 1.8 (1.0)
  Week 8 | 1.5 (1.0)
  Week 12 | 1.3 (1.0)
  Week 16 | 1.5 (1.1)
  Week 20 | 1.6 (1.1)
  Week 24 | 1.4 (1.1)

20. Secondary Outcome: PSI "Pain From Skin Lesions" Component Score at Each Visit
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 8, 12, 16, 20, and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 77
units on a scale
  Week 1: number analyzed (Participants) | 74
  Week 1 | 1.2 (1.2)
  Week 2: number analyzed (Participants) | 74
  Week 2 | 1.2 (1.1)
  Week 3: number analyzed (Participants) | 74
  Week 3 | 1.0 (1.0)
  Week 4 | 1.0 (1.0)
  Week 8 | 0.8 (0.9)
  Week 12 | 0.7 (0.9)
  Week 16 | 0.9 (1.1)
  Week 20 | 0.9 (1.1)
  Week 24 | 0.8 (1.0)

21. Secondary Outcome: Patient Assessment of Treatment Satisfaction at Week 12
Description: Participants indicated their level of satisfaction with the medication's control of psoriasis on a scale from "very dissatisfied" to "very satisfied".
Time Frame: Week 12
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 74
percentage of participants
  Very dissatisfied | 4.1 [0.8 to 11.4]
  Dissatisfied | 13.5 [6.7 to 23.5]
  Neither satisfied nor dissatisfied | 21.6 [12.9 to 32.7]
  Satisfied | 32.4 [22.0 to 44.3]
  Very satisfied | 28.4 [18.5 to 40.1]

22. Secondary Outcome: Patient Assessment of Treatment Satisfaction at Week 24
Description: as for outcome 21
Time Frame: Week 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 75
percentage of participants
  Very dissatisfied | 8.0 [3.0 to 16.6]
  Dissatisfied | 25.3 [16.0 to 36.7]
  Neither satisfied nor dissatisfied | 13.3 [6.6 to 23.2]
  Satisfied | 24.0 [14.9 to 35.3]
  Very satisfied | 29.3 [19.4 to 41.0]

23. Secondary Outcome: Percent Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Weeks 12 and 24
Description: The dermatology life quality index (DLQI) is a skin disease-specific instrument to evaluate health-related quality of life. The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answered 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is from 0 (best possible score) to 30 (worst possible score). Percent change from baseline was calculated as (Baseline Value - Post-baseline Value) / Baseline Value * 100, hence a positive value indicates improvement.
Time Frame: Baseline and weeks 12 and 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 75
percent change
  Week 12: number analyzed (Participants) | 74
  Week 12 | 53.60 (35.46)
  Week 24 | 36.95 (92.77)

24. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: From first dose of etanercept to 30 days after last dose, up to 28 weeks.
Population: Participants who received at least 1 dose of etanercept during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 80
Participants
  All adverse events (AEs) | 19
  Serious adverse events | 2
  AEs leading to discontinuation of etanercept | 2
  Fatal adverse events | 0
  Treatment-related adverse events (TRAEs) | 10
  Treatment-related serious adverse events | 1
  TRAEs leading to discontinuation of etanercept | 1
  Fatal treatment-related adverse events | 0

ADVERSE EVENTS:
Time Frame: From first dose of etanercept to 30 days after last dose, up to 28 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 2/80
Other Adverse Events (participants affected / at risk) | 18/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=80)
Injection site reaction (General disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=80)
Diarrhoea (Gastrointestinal disorders) | 1
Injection site hypersensitivity (General disorders) | 1
Injection site reaction (General disorders) | 2
Injection site swelling (General disorders) | 1
Pyrexia (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinobronchitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Injection related reaction (Injury, poisoning and procedural complications) | 2
Meniscus injury (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-02-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT02749370/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT02749370/SAP_001.pdf